CLINICAL TRIAL: NCT05604404
Title: Response of Intracranial Pressure Based on Head-of-Bed Positioning in Aneurysmal Subarachnoid Hemorrhage
Brief Title: Effects of Head-of-Bed on Intracranial Pressure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Sprague W Hazard III, Assistant Professor of Anesthesiology; Director of Neuroanesthesia, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00020509
Record Dates: First submitted 2022-10-26; First posted 2022-11-03 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
Keywords: Hemorrhage, Subarachnoid; Intracranial Pressure
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Supine Position

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Positional Changes (Experimental): The patient will begin in a supine position with the head-of-bed (HOB) at zero (0) degrees. The patient will remain in this position for five (5) minutes while pressure data is collected every fifteen (15) seconds. Next, the HOB will be adjusted to thirty (30) degrees. The patient will remain in this position for five (5) minutes while pressure data is collected every fifteen (15) seconds. Lastly, the HOB will remain at thirty (30) degrees and the foot-of-bed (FOB) will be adjusted to place the patient's leg in a dependent position. The patient will remain in this position for five (5) minutes while pressure data is collected every fifteen (15) seconds.
  Interventions: Other: Supine; Other: Semi-Recumbent; Other: Semi-Recumbent with Legs Flexed

INTERVENTIONS:
Other: Supine — The patient will be positioned supine with head-of-bed at zero degrees.
Other: Semi-Recumbent — The patient will be placed in a semi-recumbent position with head-of-bed at thirty degrees.
Other: Semi-Recumbent with Legs Flexed — The patient will be placed in a semi- recumbent position with head-of-bed at thirty degrees and legs flexed.

SUMMARY:
The purpose of this study is to evaluate how pressure inside the skull responds to position changes in patients with brain bleeds.

DETAILED DESCRIPTION:
The optimal positioning of the head-of-bed (HOB) has remained controversial in the neurosurgical field. Very limited data exists outlining the effects of HOB positioning in subarachnoid hemorrhage (SAH) patients. One study by Schulz-Stubner and Thiex assess the effects of HOB positioning in SAH and traumatic brain injury (TBI) patients. While this study offers some valuable insight into the changes in cerebral hemodynamics seen when the HOB changes, it congregates data from two very different pathologies. This could potentially misrepresent the true effects patients experience. A study by Kung et al. assesses cerebral blood flow dynamics and HOB changes in the setting of SAH but does not evaluate the effects on intracranial pressure (ICP) (Kung, et al., 2013). There appear to be no studies which evaluate the effect of HOB positioning on ICP in patients with SAH. No current data exists to determine if dependent leg positioning would help to further lower ICP. Theoretically, placing a patient's legs in a dependent position would lead to increased venous pooling of blood in the legs which might translate to lower ICP.

ELIGIBILITY:
Inclusion Criteria:

* Patients with subarachnoid hemorrhage confirmed by CT scan, MRI, or cerebral angiogram
* Age ≥ 18 years old
* Patients with intracranial pressure monitoring device
* Patients with continuous arterial blood pressure monitoring
* The subject or legally authorized representative must be available and able to consent

Exclusion Criteria:

* Intubated patients who are prone
* Patients with left ventricular ejection fraction <20% as evidenced by echocardiogram previously documented at any time in the electronic medical record
* Patients with a diagnosis of pulmonary hypertension
* Patients with a diagnosis of cirrhosis and/or evidence of liver failure. Evidence of liver failure will be assessed by the presence of ascites, edema, abnormal lab values including low albumin, elevated PTT, elevated PT, elevated INR, or elevated bilirubin without another etiology, or MELD score >8.
* Patients who are clinically unstable defined as those who are unable to lie flat for 30 minutes for any reason, patients on more than one continuous IV medications to increase blood pressure, or patients who are actively undergoing resuscitation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Intracranial Pressure Change, measured in mmHg | Measured every fifteen seconds for twenty minutes.
Cerebral Perfusion Pressure Change, measured in mmHg | Measured every fifteen seconds for twenty minutes.
Response of Intracranial Pressure to Positional Changes During Hospitalization | During hospitalization, maximum ten sequential days.
  The response of intracranial pressure to positional changes will be monitored during hospitalization.

SECONDARY OUTCOMES:
Do Patients Experiencing Vasospasm Have Similar ICP Responses to Positional Changes? | Measured once per day; for up to ten days.
  Transcranial Doppler of Middle Cerebral Artery; Mean Velocity
Do Patients Experiencing Vasospasm Have Similar ICP Responses to Positional Changes? | Measured every fifteen seconds for twenty minutes.
  Intracranial Pressure; measured in mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Cain Dudek, BS, Principal Investigator — Penn State Hershey Medical Center College of Medicine
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kung DK, Chalouhi N, Jabbour PM, Starke RM, Dumont AS, Winn HR, Howard MA 3rd, Hasan DM. Cerebral blood flow dynamics and head-of-bed changes in the setting of subarachnoid hemorrhage. Biomed Res Int. 2013;2013:640638. doi: 10.1155/2013/640638. Epub 2013 Nov 25. PMID 24371827
- [Background] Mokri B. The Monro-Kellie hypothesis: applications in CSF volume depletion. Neurology. 2001 Jun 26;56(12):1746-8. doi: 10.1212/wnl.56.12.1746. PMID 11425944
- [Background] Munakomi S, Das JM. Brain Herniation. 2023 Aug 13. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK542246/ PMID 31194403
- [Background] Prunell GF, Mathiesen T, Diemer NH, Svendgaard NA. Experimental subarachnoid hemorrhage: subarachnoid blood volume, mortality rate, neuronal death, cerebral blood flow, and perfusion pressure in three different rat models. Neurosurgery. 2003 Jan;52(1):165-75; discussion 175-6. doi: 10.1097/00006123-200301000-00022. PMID 12493115
- [Background] Suarez JI, Tarr RW, Selman WR. Aneurysmal subarachnoid hemorrhage. N Engl J Med. 2006 Jan 26;354(4):387-96. doi: 10.1056/NEJMra052732. No abstract available. PMID 16436770
- [Background] Zoerle T, Lombardo A, Colombo A, Longhi L, Zanier ER, Rampini P, Stocchetti N. Intracranial pressure after subarachnoid hemorrhage. Crit Care Med. 2015 Jan;43(1):168-76. doi: 10.1097/CCM.0000000000000670. PMID 25318385
- [Background] Schulz-Stubner S, Thiex R. Raising the head-of-bed by 30 degrees reduces ICP and improves CPP without compromising cardiac output in euvolemic patients with traumatic brain injury and subarachnoid haemorrhage: a practice audit. Eur J Anaesthesiol. 2006 Feb;23(2):177-80. doi: 10.1017/S0265021505232118. No abstract available. PMID 16426476